CLINICAL TRIAL: NCT01057511
Title: Investigation of the Differences of Progesterone Concentration in Serum and Endometrium After Administration With Vaginal and Intramuscular Progesterone
Brief Title: Compare the Difference of P4 Concentration in Serum and Endometrium After Vaginal and IM P Administration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMR200113-600
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-04

CONDITIONS: Postmenopausal Endometrium
Keywords: Crinone; progesterone; endometrial progesterone concentration
MeSH Terms: interventions — Progesterone; Inosine Monophosphate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- progesterone (Active Comparator): Each subject in this group will be give progesterone oil 20mg via intramuscular route once a day for 7 days totally
  Interventions: Drug: Progesterone
- Crinone 8% (Experimental): Each subjects in this group will be given Crinone 8% 90mg via vaginal route once a day for 7 days totally.
  Interventions: Drug: Crinone 8%

INTERVENTIONS:
Drug: Crinone 8% — Crinone 8%, 90mg / p.v. / Qd, 7 days totally.
  Other Names: progesterone vaginal gel
  Arms: Crinone 8%
Drug: Progesterone — Progesterone 20mg/ i.m./ Qd, 7 days totally.
  Other Names: IMP
  Arms: progesterone

SUMMARY:
Crinone is a micronized progesterone gel which is administrated via vaginal route and targeted drug delivery to uterine (first uterine pass effect) with lower serum concentration. This study is to investigate the difference of progesterone concentration in serum and endometrium after administration with crinone and intramuscular progesterone.

The study will be conducted as a single centre, randomized, active controlled study. Recruitment duration will be 6-8 months long. Day 1 of Crinone administration will be the baseline. On Day 7 of Crinone administration endometrial tissue will be taken for P4 test. Last visit will be at 3-5 days after withdraw bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Perimenopausal women aged <55 years old with amenorrhea>=2 months or reproductive aged women with amenorrhea >= 6months due to premature ovarian failure or other reasons.;
* Serum progesterone level < 1ng/mL
* Endometrial thickness ≥5mm
* No contraindication of progesterone administration;
* Informed consent is signed.

Exclusion Criteria:

* The other kind of progestin was applied 1 month before recruitment;
* Any serious diseases that does not allow to receive the progestin treatment;
* Under any vaginal treatment;
* Any vaginal infectious disease;
* Any other hormone treatment contraindications;
* drug abuse or untreated STD;
* Prior hypersensitivity to Crinone or one of their excipients.
* Pregnant women who indicate hCG positive.

Max Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: progesterone level in endometrium and in serum | after 7 days of progesterone therapy
  The women who singed informed consent were randomized into two groups, respectively received Crinone 90mg via vaginal route or progesterone 20mg via IM route, once per day, for seven days. After 7 days therapy, endometrium biopsy was taken via vaginal route for tissue P concentration test by radioimmunoassay method. Blood sample were drawn for serum progesterone level.

CONTACTS AND LOCATIONS:
Overall Officials: AIJUN SUN, PhD, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China